CLINICAL TRIAL: NCT02031198
Title: An 18-months Open Label Phase I Follow-up Study on Patients With Alzheimer's Disease Who Have Completed the AADvac1 Phase I Study "AXON CO 18700"
Brief Title: 18-months Safety Follow-up Study of AADvac1, an Active Tau Vaccine for Alzheimer's Disease
Acronym: FUNDAMANT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Axon Neuroscience SE (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-AD-002; 2013-004499-36 (EudraCT Number)
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; tau; dementia; elderly; cognitive; disease modifying; treatment; immunization; vaccine
MeSH Terms: conditions — Alzheimer Disease; Pick Disease of the Brain; Dementia | interventions — AADvac1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AADvac1 (Experimental): Patients who have received 6 doses in the previous trial will be administered 1-2 booster doses of AADvac1 (2 if their antibody titers decline below those achieved in the previous trial).
  Patients who have received 3 doses in the previous trial will be administered another 3 doses, then vaccinated with booster doses as above.
  Interventions: Drug: AADvac1

INTERVENTIONS:
Drug: AADvac1 — Active immunization against pathological Alzheimer's disease tau protein
  Other Names: Axon peptide 108 (coupled to KLH), 40ug/0.3mL; Axon peptide 108 conjugated to KLH

SUMMARY:
This follow-up study continues to observe patients who have completed the phase 1 trial of AADvac1, for another 18 months.

Long-term safety and behavior of the immune response to AADvac1 over time are the main points of interest.

AADvac1 is a vaccine directed against pathologically modified Alzheimer tau protein that is the main constituent of neurofibrillary tangles (NFTs), and is intended to be a disease-modifying treatment for Alzheimer's disease, i.e. to halt its progress.

As this study is a Phase I study focused on tolerability and safety, efficacy will be assessed in an exploratory manner.

DETAILED DESCRIPTION:
AADvac1 is a candidate therapeutic vaccine for Alzheimer's disease that targets misfolded tau protein, a common denominator of neurofibrillary pathology. Based on preclinical results, the intervention is expected to reduce the number of neurofibrillary tangles, remove hyperphosphorylated tau protein and reduce the amount of oligomerized and insoluble pathological tau in the brain, to halt the spread of neurofibrillary pathology through the brain, and thus prevent associated cognitive decline.

The vaccine's antigenic determinant is a synthetic peptide derived from a tau protein sequence, which is coupled to keyhole limpet hemocyanin (KLH) and uses aluminum hydroxide (Alhydrogel) as an adjuvant.

At present AADvac1 is intended as an active immunotherapy for patients with diagnosed Alzheimer's disease (AD). According to need, patients will receive additional immunization doses beyond those administered in the preceding pase 1 trial; the raised titers of therapeutic antibodies and possible benefits of the treatment can extend beyond the duration of the study.

Because of the central role of pathological misfolded tau protein in the etiology of AD, the vaccine is expected to be more effective than active or passive immunotherapies aiming to eliminate the amyloid β plaques that have been clinically investigated so far.

ELIGIBILITY:
Inclusion Criteria:

1. Completion of visit V8 of the AADvac1 phase I study AXON CO 18700 (EUDRACT 2012-003916-29).
2. Informed consent capability (as determined by an independent neurologist/psychiatrist).
3. Written informed consent signed and dated by the patient and the caregiver.
4. Availability of a partner/caregiver knowing the patient and being able to accompany the patient to the visits
5. Adequate visual and auditory abilities and language skills to allow neuropsychological testing.
6. Female patients are only eligible for the study if they are either surgically sterile or at least 2 years postmenopausal.
7. Sexually active males must be using reliable contraception methods (i.e. condoms) or be surgically sterile.

Exclusion Criteria:

1. Pregnant women.
2. Participation in another clinical trial during the course of this study.
3. Contraindication for MRI imaging such as MRI-incompatible metallic endoprosthesis or MRI-incompatible stent implantation
4. History and/or presence of autoimmune disease, if considered relevant by the investigator.
5. Significant systemic illness (e.g., chronic renal failure, chronic liver disease, poorly controlled diabetes, poorly controlled congestive heart failure, congenital long QT syndrome, other deficiencies), if considered relevant by the investigator.
6. Current treatment with immunosuppressive drugs.

Ages: 50 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-01; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Tolerability and safety profile of AADvac1 in patients with mild-to-moderate Alzheimer's disease | Tolerability & safety are assessed over a period of 18+ months
  Safety is assessed via recording of all Adverse Events and Adverse Events
  Patients are observed via:
  MRI Clinical & neuro-psychiatric observation Cognitive testing ECG Blood biochemistry, hematology, coagulation measurement Urine analysis

SECONDARY OUTCOMES:
Immunogenicity of AADvac1 | Immune response to the vaccine will be assessed over 18 month
  Measurement of:
  Titres of antibodies reactive with AADvac1 Titres of antibodies reactive with Alzheimer tau protein Antibody isotype profiles
Patient cognition | 18+ months
  Tests used:
  ADAS-Cog (Alzheimer's Disease Assessment Scale-cognitive subscale) COWAT (Controlled oral word association test) Category fluency

CONTACTS AND LOCATIONS:
Overall Officials: Reinhold Schmidt, Professor, Principal Investigator — Medizinische Universität Graz
Locations (4):
- Austria (4):
  - Univeristätsklinik für Neurologie, PMU, Christian-Doppler Klinik, Salzburg, Salzburg
  - Medizinische Universitat Graz, Graz, Styria
  - Medizinische Universitat Wien, Vienna, Vienna
  - Sozialmedizinisches Zentrum Ost (SMZ Ost) /Donauspital, Memory Clinic and Karl Landsteiner Institut for Amnestic disorders, Vienna, Vienna

REFERENCES:
- [Derived] Novak P, Schmidt R, Kontsekova E, Kovacech B, Smolek T, Katina S, Fialova L, Prcina M, Parrak V, Dal-Bianco P, Brunner M, Staffen W, Rainer M, Ondrus M, Ropele S, Smisek M, Sivak R, Zilka N, Winblad B, Novak M. FUNDAMANT: an interventional 72-week phase 1 follow-up study of AADvac1, an active immunotherapy against tau protein pathology in Alzheimer's disease. Alzheimers Res Ther. 2018 Oct 24;10(1):108. doi: 10.1186/s13195-018-0436-1. PMID 30355322
- [Derived] Novak P, Schmidt R, Kontsekova E, Zilka N, Kovacech B, Skrabana R, Vince-Kazmerova Z, Katina S, Fialova L, Prcina M, Parrak V, Dal-Bianco P, Brunner M, Staffen W, Rainer M, Ondrus M, Ropele S, Smisek M, Sivak R, Winblad B, Novak M. Safety and immunogenicity of the tau vaccine AADvac1 in patients with Alzheimer's disease: a randomised, double-blind, placebo-controlled, phase 1 trial. Lancet Neurol. 2017 Feb;16(2):123-134. doi: 10.1016/S1474-4422(16)30331-3. Epub 2016 Dec 10. PMID 27955995